CLINICAL TRIAL: NCT02652091
Title: Impact of the BETACONNECT Auto-injector on BETASERON Therapy Adherence and Patient Satisfaction
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17942
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Adherence; Persistence; Patient satisfaction
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Patient Satisfaction | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interferon beta-1b: Patients diagnosed with relapse-remitting multiple sclerosis (RRMS) or clinically isolated syndrome (CIS) who are injecting Betaseron via the Betaconnect device.
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046); Device: BETACONNECT device

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Applied via the BETACONNECT device. Dose as prescribed by physician.
Device: BETACONNECT device — Used to apply Betaseron.

SUMMARY:
The primary objective of this study is to assess adherence and persistence to BETASERON therapy in patients who are using the BETACONNECT auto-injector device (BETACONNECT device).

The secondary objective of this study is to assess patient-reported satisfaction with the BETACONNECT device.

ELIGIBILITY:
Inclusion Criteria:

* Male and females greater than or equal to 18 years of age
* Diagnosis of RRMS according to revised McDonald Criteria (2010) or (CIS)
* Prescribed BETASERON (note: decision to treat with BETASERON must be made independent of participation in this study)
* Confirmation of insurance coverage for BETASERON treatment
* Access to a personal computer to complete online patient satisfaction survey at Week 6

Exclusion Criteria:

* Currently enrolled in a clinical trial or other observational study for Multiple Sclerosis treatment
* Documented substance abuse within the previous 6 months prior to study enrollment
* Any major laboratory value abnormality that the investigator believes would preclude the patient from participating in the study
* Any medical disorder, condition or history that in the opinion of the investigator would impair the patient's ability to participate in or complete the study
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with relapse-remitting multiple sclerosis (RRMS) or clinically isolated syndrome (CIS)
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Number of BETASERON injections as captured by the BETACONNECT device | At 6 months
Time (days) between BETASERON injections as captured by BETACONNECT device | At 6 months

SECONDARY OUTCOMES:
Patient reported satisfaction by a questionnaire | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (22):
- United States (22):
  - Cullman, Alabama
  - Boca Raton, Florida
  - New Port Richey, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Fulton, Maryland
  - Foxborough, Massachusetts
  - Deckerville, Michigan
  - St Louis, Missouri
  - Stratford, New Jersey
  - Teaneck, New Jersey
  - Staten Island, New York
  - Medford, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Lititz, Pennsylvania
  - Franklin, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Lubbock, Texas
  - Round Rock, Texas
  - Fairfax, Virginia
  - Virginia Beach, Virginia